CLINICAL TRIAL: NCT00538512
Title: Comparative Study of Influenza Vaccines in Adults, FLUVACS-year 4
Acronym: FLUVACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Arnold S. Monto, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: FLUVACS
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Results first posted 2011-09-12 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Influenza
Keywords: Influenza; Live attenuated influenza vaccine; Inactivated influenza vaccine; Vaccine Efficacy
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluMist

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TIV (Active Comparator): the trivalent inactivated influenza vaccine - Fluzone, manufactured by Sanofi-Pasteur
  Interventions: Biological: Fluzone
- LAIV (Active Comparator): live-attenuated influenza vaccine Flumist, manufactured by MedImmune
  Interventions: Biological: Flumist
- Placebo (Placebo Comparator): Physiologic saline administered as a nasal spray or intramuscular injection
  Interventions: Other: Physiologic saline

INTERVENTIONS:
Biological: Fluzone — single dose licensed trivalent inactivated influenza vaccine (2007-08)
  Arms: TIV
Biological: Flumist — single dose licensed live-attenuated influenza vaccine Flumist (2007-08)
  Arms: LAIV
Other: Physiologic saline — single dose placebo administered as an intranasal spray or intramuscular injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the absolute (versus placebo) and relative (one vaccine compared to the other) efficacies of the live attenuated and inactivated influenza vaccines in preventing laboratory confirmed symptomatic influenza caused by circulating strains whether similar or dissimilar to strains included in the vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men and women
* Age 18-49 years
* Who reside geographically close to one of the four study sites in Michigan

Exclusion Criteria:

* Persons with any of the health conditions for which the inactivated vaccine is recommended
* Persons for whom either vaccine is contraindicated

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1952 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnold S. Monto, MD, Principal Investigator — University of Michigan School of Public Health
Locations (4):
- United States (4):
  - University of Michigan School of Public Heatlh, Ann Arbor, Michigan
  - Western Michigan University Health Services, Kalamazoo, Michigan
  - Central Michigan University Health Services, Mount Pleasant, Michigan
  - Eastern Michigan University Health Services, Ypsilanti, Michigan

REFERENCES:
- [Background] Ohmit SE, Victor JC, Rotthoff JR, Teich ER, Truscon RK, Baum LL, Rangarajan B, Newton DW, Boulton ML, Monto AS. Prevention of antigenically drifted influenza by inactivated and live attenuated vaccines. N Engl J Med. 2006 Dec 14;355(24):2513-22. doi: 10.1056/NEJMoa061850. PMID 17167134
- [Result] Monto AS, Ohmit SE, Petrie JG, Johnson E, Truscon R, Teich E, Rotthoff J, Boulton M, Victor JC. Comparative efficacy of inactivated and live attenuated influenza vaccines. N Engl J Med. 2009 Sep 24;361(13):1260-7. doi: 10.1056/NEJMoa0808652. PMID 19776407
- [Result] Monto AS, Petrie JG, Cross RT, Johnson E, Liu M, Zhong W, Levine M, Katz JM, Ohmit SE. Antibody to Influenza Virus Neuraminidase: An Independent Correlate of Protection. J Infect Dis. 2015 Oct 15;212(8):1191-9. doi: 10.1093/infdis/jiv195. Epub 2015 Apr 8. PMID 25858957
- [Result] Ohmit SE, Petrie JG, Cross RT, Johnson E, Monto AS. Influenza hemagglutination-inhibition antibody titer as a correlate of vaccine-induced protection. J Infect Dis. 2011 Dec 15;204(12):1879-85. doi: 10.1093/infdis/jir661. Epub 2011 Oct 12. PMID 21998477
- [Derived] Gilbert PB, Fong Y, Juraska M, Carpp LN, Monto AS, Martin ET, Petrie JG. HAI and NAI titer correlates of inactivated and live attenuated influenza vaccine efficacy. BMC Infect Dis. 2019 May 22;19(1):453. doi: 10.1186/s12879-019-4049-5. PMID 31117986
- [Derived] Petrie JG, Ohmit SE, Johnson E, Cross RT, Monto AS. Efficacy studies of influenza vaccines: effect of end points used and characteristics of vaccine failures. J Infect Dis. 2011 May 1;203(9):1309-15. doi: 10.1093/infdis/jir015. Epub 2011 Mar 4. PMID 21378375

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluzone - Trivalent Inactivated Influenza Vaccine: the trivalent inactivated influenza vaccine - Fluzone, manufactured by Sanofi-Pasteur
- Flumist - Live-attenuated Influenza Vaccine: live-attenuated influenza vaccine Flumist, manufactured by MedImmune
Period: Overall Study
Arm/Group | Fluzone - Trivalent Inactivated Influenza Vaccine | Flumist - Live-attenuated Influenza Vaccine | Placebo
Started | 814 | 813 | 325
Completed | 787 | 783 | 312
Not Completed | 27 | 30 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluzone - Trivalent Inactivated Influenza Vaccine | Flumist - Live-attenuated Influenza Vaccine | Placebo | Total
Number analyzed (Participants) | 814 | 813 | 325 | 1952
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 814 | 813 | 325 | 1952
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.2 (7.4) | 23.5 (7.7) | 22.9 (6.7) | 23.3 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 494 | 519 | 201 | 1214
  Male | 320 | 294 | 124 | 738
Region of Enrollment [Number; unit: participants]
  United States | 814 | 813 | 325 | 1952

OUTCOME MEASURES:

1. Primary Outcome: Laboratory-confirmed (Culture and/or PCR) Symptomatic Influenza
Time Frame: one influenza season - 2007-2008
Population: ITT
Measure: Number; unit: participants
Arm/Group | Fluzone - Trivalent Inactivated Influenza Vaccine | Flumist - Live-attenuated Influenza Vaccine | Placebo
Number analyzed (Participants) | 814 | 813 | 325
participants | 28 | 56 | 35

2. Secondary Outcome: Measure Immune Response Induced by the Vaccines and Identify Serologic Correlates of Immune Protection
Description: Measure immune response induced by the vaccines. Response was defined as greater than or equal to 4 fold rise in antibody titers measured by hemagglutination inhibition (HAI), microneutralization (MN), or neuraminidase inhibition (NAI) assays between sera collected at the prevaccination visit and those collected at the postvaccination visit.
Time Frame: Time between prevaccination visit and postvaccination visit; typically about 30 days.
Population: Protocol only required that a subset of all specimens be run in order to get statistically significant outcomes; because the MN assay is labor intensive a subset of sera was processed in that assay for the Flumist-live attenuated influenza vaccine group to maintain comparable tested sample sizes among the three arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone - Trivalent Inactivated Influenza Vaccine | Flumist - Live-attenuated Influenza Vaccine | Placebo
Number analyzed (Participants) | 178 | 227 | 92
Participants
  HAI assay | 137 | 48 | 92
  NAI assay | 65 | 14 | 5
  MN assay: number analyzed (Participants) | 52 | 60 | 59
  MN assay | 35 | 10 | 2

3. Secondary Outcome: Immune Response to Vaccination and Infection
Description: Response was defined as greater than or equal to 4 fold rise in antibody titers measured by hemagglutination inhibition (HAI), microneutralization (MN), or neuraminidase inhibition (NAI) assays between sera collected at the postvaccination visit and those collected at the postseason visit.
Time Frame: Postvaccination to postseason visit; typically about 3 months.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone - Trivalent Inactivated Influenza Vaccine | Flumist - Live-attenuated Influenza Vaccine | Placebo
Number analyzed (Participants) | 22 | 52 | 29
Participants
  HAI assay | 4 | 40 | 28
  NAI assay | 9 | 33 | 22
  MN assay: number analyzed (Participants) | 22 | 30 | 29
  MN assay | 6 | 20 | 26

4. Secondary Outcome: Identify Serologic Correlates of Immune Protection. Suggest Changing to: Number of Participants Demonstrating Postvaccination Seroconversion.
Description: Identify serologic correlates of immune protection. Seroconversion is defined as either prevaccination titer of less than 8 and postvaccination titer of greater than or equal to 32 or prevaccination titer of greater than or equal to 8 and greater than or equal to 4 fold rise in strain specific hemagglutination-inhibition (HAI) antibody titer between prevaccination and postvaccination sera. Data is shown separately for cases (subjects with symptomatic influenza A laboratory confirmed by isolation in cell culture or identification in real-time polymerase chain reaction (PCR) assay) and non-cases (subjects without cell culture, real time PCR or serologic evidence of influenza infection).
Time Frame: Time between prevaccination and postvaccination, typically about 30 days.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fluzone - Trivalent Inactivated Influenza Vaccine | Flumist - Live-attenuated Influenza Vaccine | Placebo
Number analyzed (Participants) | 259 | 289 | 110
Participants
  Cases: number analyzed (Participants) | 22 | 53 | 30
  Cases | 20 | 13 | 0
  Noncases: number analyzed (Participants) | 237 | 236 | 80
  Noncases | 178 | 48 | 3

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Fluzone - Trivalent Inactivated Influenza Vaccine | Flumist - Live-attenuated Influenza Vaccine | Placebo
Serious Adverse Events (participants affected / at risk) | 8/814 | 4/813 | 3/325
Other Adverse Events (participants affected / at risk) | 0/814 | 0/813 | 0/325
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluzone - Trivalent Inactivated Influenza Vaccine (N=814) | Flumist - Live-attenuated Influenza Vaccine (N=813) | Placebo (N=325)
Abdominal pain, vomiting, diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Anorexia (Gastrointestinal disorders) | 1 | 0 | 0
Appendicitis, appendectomy (Gastrointestinal disorders) | 1 | 0 | 0
Breast Cancer/Mastectomy (Reproductive system and breast disorders) | 0 | 1 | 0
Cellulitis left leg (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cervical cancer (Reproductive system and breast disorders) | 1 | 0 | 0
Cholecystitis, cholecystectomy, cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 2
Depression/anxiety (Nervous system disorders) | 0 | 0 | 1
Head injury bike accident (Surgical and medical procedures) | 1 | 0 | 0
Mononucleosis (Infections and infestations) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
surgical repair of torn ACL (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
surgury - remove tumor in left ovary/fallopian tube (Reproductive system and breast disorders) | 0 | 1 | 0
Cholecystitis, cholecystectomy, cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0
Appendectomy (Gastrointestinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No